CLINICAL TRIAL: NCT04978103
Title: Effects of Gum Arabic Supplementation on the Components of Metabolic Syndrome Among Post Menopausal Females in Khartoum State 2019
Brief Title: Effects of Gum Arabic on Metabolic Syndrome Parameters in Postmenopausal Women
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Khartoum (Other)
Collaborators: Ministry of Higher Education and Scientific Research, Republic of Sudan (Other Government)
Responsible Party: Principal Investigator, Fatima Elhaj, Principal Investigator, University of Khartoum
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMPB/0047815
Record Dates: First submitted 2021-07-10; First posted 2021-07-27 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Metabolic Syndrome in Postmenopausal Females
Keywords: Gum Arabic; Inflammatory markers; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Gum Arabic

STUDY DESIGN:
Intervention Model Description: Postmenopausal females are randomly selected to receive Gum Arabic treatment and intended outcomes will be measured before and after the intervention
Masking Description: Both the investigators and outcome assessors will be given codes of the participants for further analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Hundred postmenopausal women were enrolled and received therapeutic dose of Gum Arabic (0.5 gm/kg/day) and followed for 12 weeks then the intended outcomes will be compared before and after completion of the study
  Interventions: Drug: Gum Arabic

INTERVENTIONS:
Drug: Gum Arabic — A dietary supplement (Powdered exudates of Acacia Senegal (Gum Arabic E-414))
  Other Names: Acacia Senegal

SUMMARY:
Gum Arabic ingestion has been proved to decrease some of the inflammatory markers in some metabolic diseases that have an inflammatory background. Nevertheless, the mechanism/s by which it does so is uncertain. This study is targeting one of the postulated molecular mechanisms at genetic level that may help to understand how Gum Arabic exerts its effect .The effects of GA on Nuclear Factor Kappa Beta, P38 Mitogen Activated Protein (MAP) Kinase levels, and on the expression of inflammatory cytokines genes are going to be assessed in postmenopausal females with Metabolic Syndrome.

DETAILED DESCRIPTION:
The Metabolic syndrome (MetS) is a collection of several interconnected biochemical, clinical, and metabolic factors that directly increase the risk of atherosclerotic cardiovascular disease and Diabetes Mellitus.

Hypertension, Dyslipidemia, insulin resistance, obesity, glucose intolerance, proinflammatory and prothrombotic states are the cornerstone features defining the syndrome. Glycerol, free fatty acids (FFA), tumor necrosis factor alpha (TNFα), interleukin 6 (IL6), interleukin 1(IL-1) and Interferon Gamma (INFγ) are some of the inflammatory substances (cytokines) that are released from different cells (monocytes and adipocytes) in MetS.

Gum Arabic is found as a mixture of sodium, calcium and potassium salts of branched polysaccharides. In the colon, GA is fermented by colonic bacteria into short chain fatty acids such as butyrate, which are partially absorbed into blood.

Butyrate treatment was found to inhibit expression of cytokine mRNAs in peripheral blood monocytes (PBMC) that are stimulated by bacterial lipopolysaccharide (LPS).

In unstimulated (PBMC), a transcription factor (Nuclear Factor kappa β (NF-κB)) controls gene expression of some inflammatory cytokines; Tumor Necrosis Factor Alpha (TNF- α), IL-1 and IL-6. NF-κB was detected mainly in the cytoplasm tightly bound to an Inhibitory protein (IκB).

When those cells are stimulated by bacterial lipopolysaccharide (LPS) or by adipokines, NFκB is activated and translocates to the nucleus to start gene expression of the inflammatory cytokines. Moreover; stimulation causes degradation of IκB which releases NFκB and allows its translocation to the nucleus.

This nuclear translocation of NFκB was found to be inhibited by butyrate (a byproduct of Gum Arabic fermentation ) providing evidence that butyrate mediated reduction of proinflammatory cytokines was achieved by reducing NFκB activation.

Consequently; the postulated mechanisms by which butyrate may regulate gene expression are through inhibition of NFκB activation and IκBα degradation.

NFκB and the inflammatory cytokines: Target for therapy in inflammatory diseases, are they?

As NFκB is involved in transcriptional regulation of many cytokines genes that contributes to immune and inflammatory responses, it may be a good target for therapy also. At present, treatment of inflammatory diseases depends greatly on aminosalicylates, corticosteroids, and immune-suppressants that decrease cytokines level especially TNF.

The anti-inflammatory and immune-modulatory properties of gum Arabic, through butyrate, described previously may offer an interesting alternative therapeutic approach for inflammatory conditions.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria Females Menopause Metabolic syndrome based on Adult panel II criteria Signed/verbal consent to participate

Exclusion Criteria:

* Exclusion criteria

  1. Patients with mental or physical disability
  2. Use of corticosteroids or any other drug that affects body weight
  3. History of Gum Arabic (GA) allergy
  4. Chronicrenal or liver disease
  5. Chronocinflammatory diseases
  6. History of CVA or MI Participants will be asked to maintain their habitually daily diet and level of activity during the period of the study and to continue any previously prescribed medication.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — postmenopausal females
Enrollment: 100 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Nuclear Factor Kappa Beta concentration in nanogram/dl | 12 weeks
  Nuclear regulatory protein
P38 Mitogen activated protein kinase in nanogram/dl | 12 weeks
  Transcription regulatory protein
Inhibitory Kappa Beta protein in nanogram/dl | 12 weeks
  inhibitory protein
Tumor necrosis factor, interferon gamma and interleukin-6 in nanogram/dl | 12 weeks
  Proinflammatory cytokines
Plasminogen activated protein inhibitor1 in picogram/dl | 12 weeks
  Protein Inhibitor
Fasting Insulin in nanogram/dl | 12 weeks
  Metabolic hormone
Insulin resistance by HOMA index | 12 weeks
  Measuring cells sensitivity to insulin

SECONDARY OUTCOMES:
Fasting Blood Sugar in mg/dl | 12 weeks
  Biochemical serological markers
Lipid profile in mg/dl | 12 weeks
  Serological markers

OTHER OUTCOMES:
waist circumference in cm | 12 weeks
  Anthropometric measurement

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Elhaj, Msc, Principal Investigator — lecturer in physiology department University of Khartoum; Shaza Elawad, MSc, Principal Investigator — lecturer in physiology department University of Khartoum
Locations (1):
- University of Khartoum, Khartoum, Sudan